CLINICAL TRIAL: NCT00051116
Title: A Phase II Study of Continuous Versus Syncopated Dosing of CC-5013 for the Treatment of Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Robert Knight MD - VP Hematology, Celgene Corporation
Organization: Celgene (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MM-008
Record Dates: First submitted 2003-01-03; First posted 2003-01-07 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Revimid; CC5013; CC-5013
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CC-5013

SUMMARY:
To evaluate the response rate, response duration, and survival of patients treated with CC-5013 in a chronic dosing schedule versus a syncopated dosing schedule.

ELIGIBILITY:
* History of histologically documented multiple myeloma with relapsed or resistant disease
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of registration. Women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Signed written informed consent and willingness to meet follow-up schedule and study procedure obligations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-05; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, MD, Study Director — Celgene Corporation
Locations (1):
- Myeloma Institute University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States